CLINICAL TRIAL: NCT01364337
Title: Design and Testing Efficacy of Blood Pressure and Glucose Lowering Diet for Taiwanese Pre-/1st Staged Hypertension Patients and/or Pre-diabetes Patients
Brief Title: Blood Pressure and Glucose Lowering Diet for Taiwanese
Acronym: Taiwan_DASH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Wen-Harn Pan, Principal investigator, National Health Research Institutes, Taiwan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EC0990602-E
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DASH diet (Active Comparator)
  Interventions: Other: DASH diet
- lower carbohydrate DASH diet (Active Comparator)
  Interventions: Other: lower carbohydrate DASH diet

INTERVENTIONS:
Other: DASH diet — DASH diet: A diet rich in whole grain, fruit and vegetable, low-fat dairy products, white meat and nuts; and lower of total fat and saturated fat.
  Arms: DASH diet
Other: lower carbohydrate DASH diet — lower carbohydrate DASH diet: A DASH diet with lower carbohydrate percentage
  Arms: lower carbohydrate DASH diet

SUMMARY:
Prevalence rates of hypertension and diabetes are high in Taiwan. Little attention is given to evidence-based dietary therapy in Taiwan. Patients, after confirmed diagnosis, are mostly prescribed with medications without comprehensive instructions on dietary therapy. DASH diet has been proven to be an effective dietary approach to reduce blood pressure for hypertension patients in US. However, dietary difference and patient profiles across countries are evident. In addition, hypertensive patients are often combined with hyperglycemia. Carbohydrate burden of DASH diet may be higher than most dietitians desire. Therefore, the investigators in tend to design a Taiwanese DASH diet and a lower carbohydrate DASH diet and test their efficacy on both blood pressure and fasting glucose lowering.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-65 years, weight 50-80 kg(±5kg)
* Two blood pressure readings and fasting blood glucose measurements:

  1. fasting blood glucose of 100-125 ml/dL and not using antidiabetic medication.
  2. systolic blood pressure of 130-159 mmHg or diastolic blood pressure of 85-99 mmHg and not using antihypertensive medication.

Exclusion Criteria:

* (a) taking blood glucose lowering, antihypertensive or oral steroid medications.

  (b) history of stroke, cardiovascular disease, abnormal liver function, cancer, stomach ulcer, inflammatory bowel disease or other chronic diseases that will influence the diet of participants.

  (c) Major surgery in the past year or about to undergo major surgery.

  (d) Is the holder of a major illness card.

  (e) Takes antipsychotics.

  (f) Harmful drinker (more than 14 drinks per week)

  (g) Has food allergies or food intolerance.

  (h) Pregnant or breastfeeding.

  (i) Unwilling to cease intake of vitamin or mineral supplements or antacids containing magnesium or calcium for the duration of the study.

  (j) Other medications or physiological states influencing the absorption of nutrients.

  (k) Other individuals deemed unsuitable to participate in the intervention by their treating physician.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 4 weeks
  Baseline and per week after intervention

SECONDARY OUTCOMES:
Fasting blood glucose, fasting insulin, cholesterol, triglycerides, HDL-C and LDL-C | will be measured at 0, 2, 4, 8, 10 and 12 weeks
Urinary magnesium, potassium, sodium and creatinine | will be measured at 0, 2, 4, 8, 10 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Han Pan, Ph. D., Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- National Health Research Institutes, Miaoli County, Taiwan